CLINICAL TRIAL: NCT03460509
Title: A Randomized Double Blind Trial Comparing Reversal With Low Doses Of Sugammadex aFter Rocuronium-induced Neuromuscular Block Under General Anesthesia in Patients Undergoing Non-cardiac Surgery(TOF TRIAL)
Brief Title: Reversal With Low Doses of Sugammadex in Patients Undergoing Non-cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Tayyba Aslam, Principal investigator, The Hospital of Vestfold
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIVAA01
Record Dates: First submitted 2017-10-17; First posted 2018-03-09 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Residual Curarization; Neuromuscular Block
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Sugammadex 0 mg/kg (Placebo Comparator): Placebo NaCl 0,9%
  Interventions: Drug: Sugammadex
- Sugammadex 0,25 mg/kg (Active Comparator): Sugammadex 0.25 mg/kg IBW
  Interventions: Drug: Sugammadex
- Sugammadex 0,5 mg/kg (Active Comparator): Sugammadex 0.50 mg/kg IBW
  Interventions: Drug: Sugammadex
- Sugammadex 1mg/kg (Active Comparator): Sugammadex 1.0 mg/kg IBW
  Interventions: Drug: Sugammadex
- Sugammadex 2mg/kg (Active Comparator): Sugammadex 2 mg/kg IBW
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Dose-response

SUMMARY:
Neuromuscular blocking agents (NMBA) are among the most commonly used drugs during general anesthesia and may induce complete muscle paralysis.They are used clinically to facilitate endotracheal intubation and to optimize surgical working conditions. Incomplete recovery from non-depolarising NMBAs continues to be a common problem in modern postoperative care unit and is associated with significant risk of microaspiration and hypoventilation which leads to pulmonary complications.Recently effective reversal of neuromuscular blockade has been described by use of lower dose of sugammadex the recommended without providing adequate answer to whether the lower dose is safe enough to avoid recurrent block.

Hypotheses:

1. Administration of sugammadex 0.25 mg/kg at TOF ratio 0.3 will successfully reverse (TOF=0.9) rocuronium induced neuromuscular block within 10 min.
2. Recurrent block (TOF ratio < 0.9) does not occur after reversal with low dose sugammadex 0.25 mg/kg.

The primary objective of this trial is to assess the dose-response characteristics of sugammadex in reversing rocuronium induced neuromuscular block and to identify the minimal effective dose

Secondary objective is to assess the safety of different doses of sugammadex (recurrent block (TOF ratio < 0.9) after reversal and the occurrence of adverse reactions)

Sugammadex is a very expensive drug which limits its use i anaesthesia department. By optimising drug dosage it may have economic impact and contribute to a wider use of sugammadex to reverse neuromuscular block before extubation and thus avoid incomplete recovery. This may lead to less risk for postoperative pulmonary complications and thereby reduce morbidity and mortality after surgery.

DETAILED DESCRIPTION:
Doses of study drug will be 0 mg/kg Ideal Body Weight (IBW), 0.25 mg/kg IBW, 0.50 mg/kg IBW, 1.0 mg/kg IBW and 2.0 mg/kg IBW. TOF will be measured every 10th second until full reversal.

ELIGIBILITY:
Inclusion Criteria:

* Patient, both genders, undergoing any elective in-hospital surgical procedure under general anesthesia requiring rocuronium neuromuscular block.
* ASA I-IV
* Signed informed consent

Exclusion Criteria:

* Patient less than 18 years of age
* Patient participating in another clinical study which could interfere with TOF trial.
* Patient with neuromuscular disease
* Patient from ICU
* BMI > 30.0 kg/m2
* Patient scheduled for local or regional anesthesia only
* Patient undergoing general anesthesia without rocuronium
* Patient with hypersensitivity to NMBAs or sugammadex. Also hypersensitivity to any active substance or to any of the following excipient: Hydrochloric acid 3.7% (to adjust pH) and/or sodium hydroxide (to adjust pH) Water for injections .
* Renal dysfunction (GFR<30 mL/min/1,73m2)
* Hepatic dysfunction
* Patient who have received sugammadex in the last 24 h.
* Pregnant or breastfeeding woman. Women in childbearing age must have a negative pregnant test before inclusion.
* Bradycardia (puls <40)
* Hypotension (Systolic BP <90 mmHg)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The time from study drug administration to reaching a TOF ratio of 0.9. | 10 minutes

SECONDARY OUTCOMES:
Number of patient with reoccurrence of neuromuscular block after initial reversal to TOF ratio 0.9. | 20 minutes
Number of patients with adverse reactions in each group | until discharge - 3 days
  Adverse reactions (anaphylactic reaction, flushing, urticaria, erythematous rash, (severe) hypotension (BPsyst> 75 mmHg), tachycardia (heart rate> 120 beats/min), bradycardia (heart rate <40 beats/min), swelling of tongue, swelling of pharynx, bronchospasm)

IPD SHARING:
Plan to Share IPD: No